CLINICAL TRIAL: NCT04759443
Title: Detection of Small Fiber Neuropathy Using Skin Properties
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Peter Novak, Director, Autonomic Laboratory, Brigham and Women's Hospital
Other Study IDs: 2021P000410
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Small Fiber Neuropathy
MeSH Terms: conditions — Small Fiber Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Image processing of skin — Image processing will be used to extract skin features that correlate with loss of small skin fibers.

SUMMARY:
Small fiber neuropathy affects millions of peoples worldwide. The neuropathy is causing disabling burning pain and dysautonomia such as dizziness with standing, brain fog, fatigue, constipation, too much or too little sweating. The detection of nerve damage is complicated and not widely available; it requires either skin biopsy or specialized equipment and training. This project utilizes the mathematical processing of skin pictures for the purpose to extract the statistical features related to loss of small fibers. This approach can improve the availability of diagnosis of small fiber neuropathy.

DETAILED DESCRIPTION:
Small fiber neuropathy, including cardiovascular diabetic neuropathy, affects millions of peoples worldwide. The neuropathy is causing disabling burning pain and dysautonomia such as dizziness with standing, brain fog, fatigue, constipation, urinary problems and cold or hot intolerance. Early and accurate diagnosis of neuropathy is essential for correct treatment. Available diagnostic methods are either invasive such as skin biopsy or available only in few specialized centers. This project addresses the limited availability of small fiber neuropathy detection.

The project utilizes utilize specialized image processing of skin pictures for the purpose to extract the statistical features that are related to loss of small fibers. The accuracy of the diagnosis verified using skin biopsies.

This approach can improve the availability of diagnosis of small fiber neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age 18 year or older
* Patients that sign the informed consent form to participate in this study
* Patients completed the autonomic testing with skin biopsies

Exclusion Criteria:

* Patients with significant hairs at the legs that will cover the skin
* Any dermatological disorder that can affect the skin composition
* The use of skin lotion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with small fiber neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of image processing | 2 years
  The diagnostic accuracy of image processing will be evaluated by using the skin biopsy as a reference.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Faulkner Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No